CLINICAL TRIAL: NCT02462278
Title: A Study Measuring Core Body Temperature Using TempuRing in Women of Childbearing Age
Brief Title: Measuring Core Body Temperature Using TempuRing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prima-Temp, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PT-001
Record Dates: First submitted 2015-05-25; First posted 2015-06-04 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Fertility
Keywords: Fertility; Continuous temperature monitor; Basal Body Temperature; Natural family planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TempuRing (Experimental): Women will wear the continuous temperature sensor, TempuRing, for 3 menstrual cycles.
  Interventions: Device: TempuRing

INTERVENTIONS:
Device: TempuRing
  Other Names: continuous temperature sensor

SUMMARY:
This study evaluates the safety and usability of a continuous temperature sensor for women. Data will compare the date of ovulation identified by the continuous temperature sensor to that of transvaginal ultrasound and serum progesterone levels. Subjects will also compare sensor results to once-daily oral temperatures and urine luteinizing hormone (LH) status.

DETAILED DESCRIPTION:
Up to 25 healthy female volunteers or females currently trying to conceive will wear the continuous temperature sensor for 3 menstrual cycles. Subjects will record their daily oral temperature, and record their urine luteinizing hormone (LH) status via ovulation prediction kits. Subjects will return to the clinic after a positive urinary LH test to receive transvaginal ultrasound scans to confirm ovulation (ultrasounds will be repeated daily until evidence of ovulation is documented by follicular collapse). Ovulation will also be confirmed by serum progesterone. Subjects will complete an online questionnaire to assess the usability and comfort of the continuous temperature monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation
2. Females aged 21 to 43 years
3. Have a body mass index (BMI) above 19 and below 29
4. Regular menstrual cycles, i.e. no greater than 7 days difference between the shortest and longest cycle in the last 6 months
5. Minimum menstrual cycle 24 days
6. Maximum menstrual cycle 35 days
7. Normal pap smear within the last year
8. Willing to use the fertility device for at least 3 cycles
9. Willing to fill in online questionnaires
10. Willing to attend clinic up to 6 times per cycle for transvaginal ultrasound and blood tests
11. Willing to perform LH urine tests at home twice a day from day 8 of cycle until it is positive
12. Willing to document the last day of the previous menses and first day of the following menses.
13. Willing to measure and record oral at the same time each morning.
14. Normal pelvic ultrasound and blood results obtained during screening tests

Exclusion Criteria:

1. Any diagnosed systemic illnesses including thyroid disease, diabetes, yeast infection, Chlamydia, gonorrhea, trichomonas, bacterial vaginosis, inflammatory diseases, or are in an immuncompromised state
2. Polycystic ovary disease
3. Endometriosis or other chronic pelvic pain or pelvic pathology
4. Taking steroid medication, including oral contraceptives or anti inflammatory drugs
5. Pregnant

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Safety of TempuRing continuous temperature monitor device in women (incidence of adverse events) | Up to 3 months
  Safety is evaluated by incidence of adverse events judged to be related to the device.

SECONDARY OUTCOMES:
Acceptability and satisfaction questionnaire to assess the usability of TempuRing | Up to 3 months
  Patients will complete an online questionnaire to assess the usability and comfort of the continuous temperature monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Costantini, PhD, Study Director — Prima-Temp, Inc
Locations (2):
- United States (2):
  - Partners HealthCare Connected Health, Boston, Massachusetts
  - University of Washington Medical Center, Seattle, Washington